CLINICAL TRIAL: NCT06204913
Title: Restaurant Menu Study: Label Noticeability
Brief Title: Menu Label Noticeability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Jennifer Falbe, Associate Professor, University of California, Davis
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1641776-1
Record Dates: First submitted 2023-11-27; First posted 2024-01-12 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2023-10

CONDITIONS: Noticing Nutrition Information; Recalling Nutrition Information

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (24):
- Left, black, icon only, 100% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the left of the item, colored black, icon only design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Left, black, icon plus text, 100% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the left of the item, colored black, icon plus text design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Left, black, boxed icon, 100% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the left of the item, colored black, boxed icon design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Right, black, icon only, 100% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the right of the item, colored black, icon only design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Right, black, icon plus text, 100% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the right of the item, colored black, icon plus text design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Right, black, boxed icon, 100% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the right of the item, colored black, boxed icon design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Left, red, icon only, 100% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the left of the item, colored red, icon only design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Left, red, icon plus text, 100% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the left of the item, colored red, icon plus text design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Left, red, boxed icon, 100% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the left of the item, colored red, boxed icon design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Right, red, icon only, 100% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the right of the item, colored red, icon only design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Right, red, icon plus text, 100% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the right of the item, colored red, icon plus text design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Right, red, boxed icon, 100% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the right of the item, colored red, boxed icon design, and height that is 100% of size of the menu text height.
  Interventions: Other: Menu label
- Left, black, icon only, 150% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the left of the item, colored black, icon only design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Left, black, icon plus text, 150% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the left of the item, colored black, icon plus text design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Right, black, icon only, 150% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the right of the item, colored black, icon only design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Right, black, icon plus text, 150% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the right of the item, colored black, icon plus text design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Left, red, icon only, 150% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the left of the item, colored red, icon only design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Left, red, icon plus text, 150% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the left of the item, colored red, icon plus text design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Right, red, icon only, 150% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the right of the item, colored red, icon only design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Right, red, icon plus text, 150% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the right of the item, colored red, icon plus text design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Left, red, boxed icon, 150% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the left of the item, colored red, boxed icon design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Left, black, boxed icon, 150% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the left of the item, colored black, boxed icon design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Right, red, boxed icon, 150% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the right of the item, colored red, boxed icon design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label
- Right, black, boxed icon, 150% height (Experimental): Participant will order meals from two menus containing labels next to items high in added sugars (exceeding half the daily value). The label will be on the right of the item, colored black, boxed icon design, and height that is 150% of size of the menu text height.
  Interventions: Other: Menu label

INTERVENTIONS:
Other: Menu label — Participants will select food items from two restaurant menus, displayed with labels as specified by their assigned group

SUMMARY:
To assess the relative noticeability of the following added-sugar menu label elements using a factorial experiment: label type (icon-only vs. icon-plus-text label vs. boxed icon), color (black vs. red), size (100% vs. 150% of the height of the menu item text), and placement (left vs. right side of item).

DETAILED DESCRIPTION:
The objective of this aim is to assess the relative noticeability of legally-viable added-sugar menu label characteristics. The investigators will use a between-subject experiment with a factorial design. Participants will be randomized to label type (icon-only vs. icon-plus-text label vs. boxed icon), color (black vs. red), size (100% vs. 150% of the height of the menu item text), and placement (left vs. right side of item). This results in 24 arms of the experiment.

The primary outcomes are noticing a nutrition label and recognition of the label. Secondary outcomes are knowledge of items that are high in added sugar and perceived message effectiveness (PME) of labels.

For dichotomous outcomes (e.g., noticing the label, recalling label meaning), the investigators will directly estimate the probability ratio using Poisson regression with a robust error variance, regressing the outcome on an indicator for the level of the factor. For continuous outcomes (e.g., knowledge, PME scale), the investigators will use linear regression models regressing the outcome on an indicator for experimental condition.

A critical alpha 0.05 will be used, and statistical tests will be two-tailed. Exploratory outcomes include selection of ≥1 item high in added sugar and grams of sugar ordered from each menu, analyzed using the methods described above. The investigators will also explore proportions or means for the following process measures about reactions to the warning labels: Perception that the labels grabbed attention and support for an added sugars warning label policy. Additionally, the investigators will explore differences in the primary outcomes between each of the 24 unique conditions. If there is evidence of interactions between label elements, investigators will modify the modeling approach to account for those interactions (e.g., using interaction terms and stratified models).The investigators will use multiple testing corrections for families of outcomes (primary and secondary).

ELIGIBILITY:
Inclusion Criteria:

* Equal or greater than 18 years of age-
* Less than 100 years of age
* English-speaking
* U.S. residents
* Participants will reflect the U.S. Census Bureau's 2021 American Community Survey 5-year estimates for gender, race/ethnicity, educational attainment, and age

Exclusion Criteria:

* Failing the attention check question
* Completing the survey in less than 33% of the median completion time

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4581 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Noticing and recall of added-sugar nutrient label - dichotomous variable "Correct" (Answered "Yes" to noticing, answered "Added sugars" to recall, and answered "high" for high low recall question) or "Incorrect" (otherwise) | up to approximately 1 minute
  Noticing a nutrition label - Measured with "Think back to the beginning of this survey when you imagined you were ordering dinner from restaurant menus. Did you notice any nutrition labels (other than the calories) next to any of the menu items?" Response options are "Yes", "No", and "Don't know".
  Recalling the label's meaning - [If answered "Yes"] Measured with "What did the nutrition label tell you about?" Response options are (displayed in survey in a random order) "Sodium", "Added sugars", "Trans fats", "Fiber", "Calcium", "Healthy items", "Unhealthy items", "Vegetarian", "Organic", "Gluten-free", "Sustainable", "None of these", "Not sure".
  High/low - [If answered "Added sugars"] "What did the label tell you about added sugars?" Response options are "High in added sugars", "Low in added sugars", "Something else", "I don't know".
  There is no formal name for this measure/scale.
Recognition of label - dichotomous variable "Correct" (selected the label they were assigned to" or "Incorrect" (any other option). | up to approximately 1 minute
  Measured with "Please look at the following labels and select which label (if any) you saw on the menus while selecting your food and beverage items." Response options will include images of 7 labels with the designs based on the participant's assigned color (black vs red) and label type (icon-only vs. boxed-icon vs, boxed icon-plus-text label) and the options, "Not sure" and "None of these".
  There is no formal name for this measure/scale. It was developed for this study.

SECONDARY OUTCOMES:
Knowledge of menu items high in added sugar - continuous variable using the percent of 8 items correctly classified | up to approximately 2 minutes
  Measured with "(While viewing menu excerpt) Click on the menu items that you think have more than half the daily limit for added sugars." Higher percents of items correctly classified represent more knowledge.
Perceived Message Effectiveness of label - continuous variable based on a 3-item scale in which each item uses a 1-5 response scale | up to approximately 2 minutes
  Measured with 3-item University of North Carolina Perceived Message Effectiveness Scale: "How much does this label make you concerned about the health effects of consuming menu items high in added sugars?", "How much does this label makes consuming menu items high in added sugars seem unpleasant?", and "How much does this label discourage you from wanting to consume menu items high in added sugars?". Response options include a 1-5 scale where higher values represent higher amounts of the construct.

OTHER OUTCOMES:
Selection of at least one item high in added sugar | up to approximately 2 minutes
  Exploratory outcome, dichotomous - "Yes" (ordered at least one item high in added sugar) or "No" (did not order any items high in added sugar), analyzed using Poisson regression to examine differences between factor levels
Grams of sugar ordered | up to approximately 2 minutes
  Exploratory outcome, continuous - total grams of sugar in menu items selected, analyzed using linear regression to examine differences between factor levels
Perception that the labels grabbed attention | up to approximately 1 minute
  Exploratory outcome, continuous - 1-5 Likert scale, descriptive analysis of proportions and means to examine differences between factor levels
Support for an added sugars warning label policy | up to approximately 1 minute
  Exploratory outcome, continuous - 1-5 Likert scale, descriptive analysis of proportions and means to examine differences between factor levels

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Falbe, ScD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No